CLINICAL TRIAL: NCT04914858
Title: The Effect of Education Given to Prospective Fathers on Daily Care of the Baby and Father-Infant Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Collaborators: Cukurova University (Other)
Responsible Party: Principal Investigator, Mustafa Kara, Kahramanmaras Sutcu Imam University, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Cukurova University
Record Dates: First submitted 2021-05-15; First posted 2021-06-07 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Pathernal Attachment; Effect of Education to Pathernal Attachment
Keywords: pathernal attachment; baby; father
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental): Education
  Interventions: Other: Education
- Control group (No Intervention): No Intervention

INTERVENTIONS:
Other: Education — Its validity and reliability is a reliable scale in Turkey
  Arms: Education group

SUMMARY:
I am conducting an experimental study examining the bonding between father and baby.

DETAILED DESCRIPTION:
The experimental group and the control group (1st group and 2nd group) will be formed by randomly selecting the spouses of women who applied to Afşin State Hospital and Elbistan State Hospital Gynecology Polyclinic. Fathers in the first group will be met face-to-face with powerpoints and visuals, and training will be provided. It is planned to provide a total of 3 educations by contacting fathers at the time of birth and 2 months after birth. The scope of the 1st education is planned to be about attachment, father-infant attachment, the benefits of father-infant attachment to the baby and the father and how this bond can be strengthened. Care and feeding of the baby is planned within the scope of the second education. In the third education, it is planned to inform the father about spending quality time with the baby and its importance. As a result, the first education will be focused on more about attachment and its importance, the second education will focus on the importance of the father's participation in the care of the baby and the information about care, and the last education the importance of the father's taking care of the baby and spending time with him. Fathers in the second group will be given a training brochure at the end of the 6th month, after the scale is applied. If the baby's health is affected by possible adverse events at birth, that father will be excluded from the study. After the birth with the fathers, when the baby reaches 6-12 months, face-to-face or phone calls will be applied and the father-infant attachment status will be analyzed by statistical analysis. The study will be done as pre-test and post-test. Güleç D. and Kavlak O. examined the validity of the father-infant Attachment Scale in Turkish society, and they came up with a questionnaire consisting of 19 questions in total.

Detail added (15.06.2021): Power analysis was performed with the study from 5 control groups from 5 experimental groups. A total of 58 workers, consisting of 29 experimental and 29 control groups, were found sufficient for the study

ELIGIBILITY:
Inclusion Criteria:

* Spouse must be in the 3rd trimester of pregnancy
* Father should be father for the first time
* The family must be a citizen of the Republic of Turkey,
* The father's education level must be at least high school and its equivalent.
* Father's age should be between 18-40.
* Father has to have a job (Active employment).

Exclusion Criteria:

* Baby must be healthy
* Parents do not have any psychological problems,

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — I am working with fathers
Enrollment: 81 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Is Education of Daily Care of the Baby and Father-Infant Attachment effective? | About 6 months per a participant
  Validity and reliability in Turkey will be made questionnaire(Pre-test, Post-test),
  ***In the study, item 16 was removed from the scale after further analysis.
  Evaluations are made as stated below:
  Items 1, 2 and 3 in the scale are coded as a=1, b= 2, c=3, d=4 and e= 5 points. Items 4. 5. 10. 12. and 14. are reverse coded as a=5, b= 4, c=3, d=2 and e=1. Items 6, 17, 18 and 19 are coded as a=1, b= 2.3, c=3.6, d=5. Items 7. 9. 11. ve 15 are reverse coded as a=5, b=3.6, c=2.3, d=1. 8th item is coded as a=5 b=1 13th item is coded as a=5, b=3, c=1

CONTACTS AND LOCATIONS:
Locations (1):
- Afsin Saglık Yuksekokulu, Afşin, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided